CLINICAL TRIAL: NCT00494507
Title: Dichlorphenamide vs. Placebo for Periodic Paralysis
Brief Title: Hyper- and Hypokalemic Periodic Paralysis Study
Acronym: HYP-HOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Robert Griggs, MD, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS045686-02 (NIH); CRC (Other: NINDS)
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Hyperkalemic Periodic Paralysis; Hypokalemic Periodic Paralysis
Keywords: periodic paralysis; dichlorphenamide
MeSH Terms: conditions — Paralysis, Hyperkalemic Periodic; Hypokalemic Periodic Paralysis | interventions — Dichlorphenamide; Double-Blind Method

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HYP Dichlorphenamide (Active Comparator): Hyperkalemic participants were randomized to Dichlorphenamide for a 9 week double-blind phase. All participants then received Dichlorphenamide for a 52 week open-label phase.
  Interventions: Drug: Dichlorphenamide (double-blind); Drug: Dichlorphenamide (open-label)
- HYP Placebo (Placebo Comparator): Hyperkalemic participants were randomized to Placebo for a 9 week double-blind phase. All participants then received Dichlorphenamide for a 52 week open-label phase.
  Interventions: Drug: Placebo (double-blind); Drug: Dichlorphenamide (open-label)
- HOP Dichlorphenamide (Active Comparator): Hypokalemic participants were randomized to Dichlorphenamide for a 9 week double-blind phase. All participants then received Dichlorphenamide for a 52 week open-label phase.
  Interventions: Drug: Dichlorphenamide (double-blind); Drug: Dichlorphenamide (open-label)
- HOP Placebo (Placebo Comparator): Hypokalemic participants were randomized to Placebo for a 9 week double-blind phase. All participants then received Dichlorphenamide for a 52 week open-label phase.
  Interventions: Drug: Placebo (double-blind); Drug: Dichlorphenamide (open-label)

INTERVENTIONS:
Drug: Dichlorphenamide (double-blind) — 50mg tablet; maximum dosage 400mg/day
  Other Names: Daranide
  Arms: HOP Dichlorphenamide; HYP Dichlorphenamide
Drug: Placebo (double-blind) — Inactive substance manufactured to look like Dichlorphenamide 50mg tablet
  Arms: HOP Placebo; HYP Placebo
Drug: Dichlorphenamide (open-label) — 50mg tablet; maximum dosage 400mg/day
  Other Names: Daranide

SUMMARY:
The purpose of this study is to compare Dichlorphenamide with placebo (an inactive substance) for prevention of episodes and for improvement of strength in hyperkalemic (HYP) and hypokalemic (HOP) periodic paralysis. This study will also look at the long-term effects of Dichlorphenamide in periodic paralysis.

DETAILED DESCRIPTION:
Periodic paralysis is a relatively rare, life-long disorder characterized by intermittent bouts of paralysis, progressive weakness, and diminished quality of life. Two drugs, acetazolamide (ACZ) and dichlorphenamide, have been prescribed to treat the disorder, however, dichlorphenamide is no longer available.

In this multi-center, parallel, randomized trial researchers will compare the effects of dichlorphenamide vs. placebo in patients with hyperkalemic (HYP) and hypokalemic (HOP) periodic paralysis.

The trial consists of two 9-week studies-one study will enroll persons with hyperkalemic periodic paralysis and the other study will enroll persons with hypokalemic periodic paralysis. Participants will be randomly assigned to one of two treatment groups: dichlorphenamide or placebo (an inactive substance). During the studies, participants will be asked to keep a daily diary to record the time, length, and severity of each episode of weakness (attack). The study coordinator will contact participants weekly to review the diary information.

The 9-week phase will be followed by a 1-year open-label dichlorphenamide extension without placebo to determine the long-term effects of dichlorphenamide on the course of the disease and on inter-attack weakness.

Duration of the trial for participants is approximately 65 weeks, including a screening phase to determine eligibility, the first 9-week treatment phase, and the one-year open-label extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Genetically definite, clinically definite or clinically probable Hyperkalemic or Hypokalemic Periodic Paralysis as outlined in the protocol
* Male and female participants, age 18 and older who are able to comply with the study conditions.
* Participants who have distinct regular episodes of weakness with an average frequency of > or = to 1 a week and < or = to 3 a day either on or off treatment, whichever is higher
* Normal thyroid-stimulating hormone (TSH) level

Exclusion Criteria:

* Evidence for Andersen-Tawil syndrome (any one of the following 3 criteria)

  1. Prolonged QT interval or complex ventricular ectopy between attacks
  2. Distinctive physical features (2 of the following 5)

     1. Low set ears
     2. Short stature
     3. Hypo-/micrognathia
     4. Clinodactyly
     5. Hypo-/hypertelorism
  3. KIR 2.1 gene mutation
* Coincidental renal, hepatic, active thyroid disease, restrictive or obstructive lung disease, other neuromuscular disease, or heart disease
* Chronic, non-congestive, angle-closure glaucoma
* Use of any of the following medications for reasons other than treatment of periodic paralysis: diuretics, antiarrhythmics, corticosteroids, beta-blockers, calcium channel blockers, antiepileptics, magnesium
* History of life-threatening episodes of respiratory muscle weakness or cardiac arrhythmias during attacks
* Pregnancy
* Known mutation in the alpha subunit of the sodium channel gene in hypokalemic periodic paralysis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-06; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Griggs, M.D., Principal Investigator — University of Rochester; Rabi Tawil, M.D., Principal Investigator — Co-Principal Investigator, University of Rochester; Michael McDermott, Ph.D. — Biostatistician, University of Rochester
Locations (12):
- United States (10):
  - UCLA Neurology, Los Angeles, California
  - University of California-San Francisco, San Francisco, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - University of Texas Southwestern-Dallas, Dallas, Texas
- University of Milan, San Donato, Milan, Italy
- Institute of Neurology-Queen's Square, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original trial design included an Acetazolamide (ACZ) drug arm which was subsequently removed. Five participants randomized to ACZ and one ineligible participant are not included in the trial results reported here.
Period: Double-Blind Phase
Arm/Group | HYP Dichlorphenamide | HYP Placebo | HOP Dichlorphenamide | HOP Placebo
Started | 12 | 9 | 24 | 20
Reached Endpoint of Acute Worsening | 0 | 2 | 0 | 5
Completed | 9 | 9 | 22 | 19
Not Completed | 3 | 0 | 2 | 1
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Subject Non-compliance | 0 | 0 | 1 | 0
Not completed — Negative DNA test | 0 | 0 | 0 | 1
Period: Open-Label Phase
Arm/Group | HYP Dichlorphenamide | HYP Placebo | HOP Dichlorphenamide | HOP Placebo
Started | 9 | 8 (1 subject randomized to Acetazolamide in this phase is not included-drug arm was removed from trial.) | 22 | 19
Completed | 9 | 7 | 17 | 14
Not Completed | 0 | 1 | 5 | 5
Not completed — Adverse Event | 0 | 1 | 5 | 3
Not completed — Worsening Disease | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HYP Dichlorphenamide | HYP Placebo | HOP Dichlorphenamide | HOP Placebo | Total
Number analyzed (Participants) | 12 | 9 | 24 | 20 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.3) | 45.2 (17.7) | 44.8 (14.6) | 44.0 (15.6) | 44.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 8 | 4 | 24
  Male | 6 | 3 | 16 | 16 | 41

OUTCOME MEASURES:

1. Primary Outcome: HYP Attack Rate
Description: The number of distinct attacks per week over the final 8 weeks (Weeks 2-9) of the double-blind treatment period as self-reported by HYP participants.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: attacks per week
Groups:
- HYP Dichlorphenamide: Hyperkalemic participants randomized to Dichlorphenamide for a 9 week double-blind phase. Dichlorphenamide (double-blind): 50mg tablet; maximum dosage 400mg/day.
- HYP Placebo: Hyperkalemic participants randomized to Placebo for a 9 week double-blind phase. Placebo (double-blind): Inactive substance manufactured to look like Dichlorphenamide 50mg tablet.
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 12 | 9
attacks per week | 0.9 [0.4 to 1.5] | 4.8 [0.5 to 7.1]

2. Primary Outcome: HOP Attack Rate
Description: The number of distinct attacks per week over the final 8 weeks (Weeks 2-9) of the double-blind treatment period as self-reported by HOP participants.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: attacks per week
Groups:
- HOP Dichlorphenamide: Hypokalemic participants randomized to Dichlorphenamide for a 9 week double-blind phase. Dichlorphenamide (double-blind): 50mg tablet; maximum dosage 400mg/day.
- HOP Placebo: Hypokalemic participants randomized to Placebo for a 9 week double-blind phase. Placebo (double-blind): Inactive substance manufactured to look like Dichlorphenamide 50mg tablet.
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 24 | 20
attacks per week | 0.3 [0.1 to 1.6] | 2.4 [0.5 to NA] — The upper quartile for the placebo group could not be calculated because more than 25% of placebo-treated subjects reached the endpoint of acute worsening.

3. Secondary Outcome: HYP Severity-weighted Attack Rate
Description: HYP participant severity-weighted attack rate is defined as the sum of average attack severity across all distinct attacks over the final 8 weeks (Weeks 2-9) of the double-blind treatment period divided by the number of weeks that the subject was followed. Attack severity (scored as 1-10 with increasing severity) is self-reported.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: severity-weighted attacks per week
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 12 | 9
severity-weighted attacks per week | 1.0 [0.4 to 2.9] | 5.8 [1.4 to 28.0]

4. Secondary Outcome: HOP Severity-weighted Attack Rate
Description: HOP participant severity-weighted attack rate is defined as the sum of average attack severity across all distinct attacks over the final 8 weeks (Weeks 2-9) of the double-blind treatment period divided by the number of weeks that the subject was followed. Attack severity (scored as 1-10 with increasing severity) is self-reported.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: severity-weighted attacks per week
Groups:
- HOP Dichlorphenamide: Hypokalemic participants were randomized to Dichlorphenamide for a 9 week double-blind phase. Dichlorphenamide (double-blind): 50mg tablet; maximum dosage 400mg/day.
- HOP Placebo: Hypokalemic participants were randomized to Placebo for a 9 week double-blind phase. Placebo (double-blind): Inactive substance manufactured to look like Dichlorphenamide 50mg tablet.
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 24 | 20
severity-weighted attacks per week | 0.6 [0.2 to 3.9] | 5.7 [1.2 to NA] — The upper quartile for the placebo group could not be calculated because more than 25% of placebo-treated subjects reached the endpoint of acute worsening and thus were assigned an arbitrarily large attack duration for purposes of analysis.

5. Secondary Outcome: HYP Attack Duration
Description: HYP participant total attack duration per week, defined as the sum of attack durations across all distinct attacks over the final 8 weeks (Weeks 2-9) of the double-blind treatment period divided by the number of weeks that the subject was followed.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: hours per week
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 12 | 9
hours per week | 10.5 [2.5 to 21.3] | 39.4 [6.2 to 139.4]

6. Secondary Outcome: HOP Attack Duration
Description: HOP participant total attack duration per week, defined as the sum of attack durations across all distinct attacks over the final 8 weeks (Weeks 2-9) of the double-blind treatment period divided by the number of weeks that the subject was followed.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: hours per week
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 24 | 20
hours per week | 2.7 [0.4 to 13.4] | 26.2 [4.0 to NA] — The upper quartile for the placebo group could not be calculated because more than 25% of placebo-treated subjects reached the endpoint of acute worsening and thus were assigned an arbitrarily large attack duration for purposes of analysis.

7. Secondary Outcome: HYP Endpoint of Acute Worsening
Description: Increase in attack frequency or severity in HYP participants necessitating withdrawal from the initial nine-week double-blind treatment period and moving directly into the open-label phase.
Time Frame: 0-9 weeks
Measure: Number; unit: participants
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 12 | 9
participants | 0 | 2

8. Secondary Outcome: HOP Endpoint of Acute Worsening
Description: Increase in attack frequency or severity in HOP participants necessitating withdrawal from the initial nine-week double-blind treatment period and moving directly into the open-label phase.
Time Frame: 0-9 weeks
Measure: Number; unit: participants
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 24 | 20
participants | 0 | 5

9. Secondary Outcome: HYP Change From Baseline to Week 9 in Average Manual Muscle Testing (MMT) Score
Description: The strength of each of 26 individual muscles was graded using a modified 13-point Medical Research Council scale ranging from 0-5. Recorded grades were converted to numerical values as follows prior to averaging across muscles to form a composite score: 0 = 0; 1 = 1; 2- = 1.67; 2 = 2; 2+ = 2.33; 3- = 2.67; 3 = 3; 3+ = 3.33; 4- = 3.67; 4 = 4; 4+ = 4.33; 5- = 4.67; 5 = 5. A higher score represents a better outcome, i.e. 5 = normal strength.
  The following muscles were tested: shoulder abductor (left/right), elbow extensor (left/right), elbow flexor (left/right), wrist extensor (left/right), wrist flexor (left/right), hip flexor (left/right), hip extensor (left/right), hip abductor (left/right), knee extensor (left/right), knee flexor (left/right), ankle dorsiflexor (left/right), ankle plantar flexor (left/right), neck extensor, neck flexor.
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 11 | 8
units on a scale | 0.13 (0.26) | 0.00 (0.16)

10. Secondary Outcome: HOP Change From Baseline to Week 9 in Average Manual Muscle Testing (MMT) Score
Description: as for outcome 9
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 23 | 17
units on a scale | 0.05 (0.21) | -0.08 (0.15)

11. Secondary Outcome: HYP Change From Baseline to Week 9 in Average Maximum Voluntary Isometric Contraction Testing (MVICT) Scores
Description: The strength of each of 10 muscles was measured using quantitative myometry and expressed as the number of standard deviations from normal (Z-score) given the participant's age, gender, and height. The scores were averaged across muscles to form a composite MVICT score: average standardized MVICT score. A positive Z-score indicates a better outcome.
  The following muscles were tested: elbow extensor (left/right), elbow flexor (left/right), knee extensor (left/right), knee flexor (left/right), and hand grip (left/right).
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 10 | 5
Z-score | 0.78 (0.52) | 0.55 (0.76)

12. Secondary Outcome: HOP Change From Baseline to Week 9 in Average Maximum Voluntary Isometric Contraction Testing (MVICT) Scores
Description: as for outcome 11
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 21 | 15
Z-score | -0.08 (0.92) | -0.27 (0.58)

13. Secondary Outcome: HYP Change From Baseline to Week 9 in Average Maximum Voluntary Isometric Contraction Testing Percent of Predicted Normal
Description: The strength of each of 10 muscles was measured using quantitative myometry and expressed as the percent of predicted normal given the participant's age, gender, and height. The scores were averaged across muscles to form a composite MVICT score: average percent of predicted normal score. A higher number indicates a better outcome.
  The following muscles were tested: elbow extensor (left/right), elbow flexor (left/right), knee extensor (left/right), knee flexor (left/right), and hand grip (left/right).
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: average percent of predicted normal
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 10 | 5
average percent of predicted normal | 10.84 (8.27) | 10.17 (14.54)

14. Secondary Outcome: HOP Change From Baseline to Week 9 in Average Maximum Voluntary Isometric Contraction Testing Percent of Predicted Normal
Description: as for outcome 13
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: average percent of predicted normal
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 21 | 15
average percent of predicted normal | -0.81 (11.27) | -2.94 (7.20)

15. Secondary Outcome: HYP Change From Baseline to Week 9 in Lean Body Mass
Description: Lean body mass was measured by dual-energy X-ray absorptiometry (DEXA).
Time Frame: Baseline and 9 weeks
Population: Participants who had lean body mass data available at baseline and week 9.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 9 | 6
kg | -1.31 (1.94) | -1.52 (1.47)

16. Secondary Outcome: HOP Change From Baseline to Week 9 in Lean Body Mass
Description: Lean body mass was measured by dual-energy X-ray absorptiometry (DEXA).
Time Frame: Baseline and 9 weeks
Population: Participants who had lean body mass data available at baseline and week 9.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 22 | 15
kg | -0.78 (1.65) | 0.44 (2.39)

17. Secondary Outcome: HYP Change From Baseline to Week 9 in SF-36 Physical Component Summary Score
Description: The Medical Outcomes Study Short Form (SF-36) questionnaire is a widely used profile measure of generic health-related quality of life. The 36 questions are allocated to eight scales: physical function (PF), physical role (RP), bodily pain (BP), general health perceptions (GH), vitality (VT), social function (SF), mental health (MH), and emotional role (RE). The physical component summary score is calculated from the four scales of PF, RP,BP, and GH. Scores are constructed as a T-score with a mean of 50 and standard deviation of 10 and no minimum or maximum score. Higher scores are associated with better quality of life.
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 12 | 8
T-score | 3.16 (7.84) | -0.11 (7.82)

18. Secondary Outcome: HOP Change From Baseline to Week 9 in SF-36 Physical Component Summary Score
Description: The Medical Outcomes Study Short Form (SF-36) questionnaire is a widely used profile measure of generic health-related quality of life. The 36 questions are allocated to eight scales: physical function (PF), physical role (RP), bodily pain (BP), general health perceptions (GH), vitality (VT), social function (SF), mental health (MH), and emotional role (RE). The physical component summary score is calculated from the four scales of PF, RP, BP, and GH. Scores are constructed as a T-score with a mean of 50 and standard deviation of 10 and no minimum or maximum score. Higher scores are associated with better quality of life.
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 20 | 17
T-score | 4.83 (7.23) | -3.75 (10.61)

19. Secondary Outcome: HYP Change From Baseline to Week 9 in SF-36 Mental Health Component Summary Score
Description: The Medical Outcomes Study Short Form (SF-36) questionnaire is a widely used profile measure of generic health-related quality of life. The 36 questions are allocated to eight scales: physical function (PF), physical role (RP), bodily pain (BP), general health perceptions (GH), vitality (VT), social function (SF), mental health (MH), and emotional role (RE). The mental health component summary score is calculated from the four scales of VT, SF, MH, and RE. Scores are constructed as a T-score with a mean of 50 and standard deviation of 10 and no minimum or maximum score. Higher scores are associated with better quality of life.
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | HYP Dichlorphenamide | HYP Placebo
Number analyzed (Participants) | 12 | 8
T-score | -3.77 (14.09) | 2.65 (8.64)

20. Secondary Outcome: HOP Change From Baseline to Week 9 in SF-36 Mental Health Component Summary Score
Description: as for outcome 19
Time Frame: Baseline and 9 weeks
Population: Participants with evaluable data at both timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | HOP Dichlorphenamide | HOP Placebo
Number analyzed (Participants) | 20 | 17
T-score | -1.10 (9.93) | -5.65 (12.58)

ADVERSE EVENTS:
Description: Adverse events were assessed via weekly phone calls with participants and at all study visits.
  One HOP participant inadvertently remained on placebo during the open-label phase and therefore is not reported in the Other Adverse Events for the HOP Open-Label Dichlorphenamide group.
Groups:
- HYP Double-Blind Dichlorphenamide: Hyperkalemic participants were randomized to Dichlorphenamide for the 9 week double-blind phase.
- HYP Double-Blind Placebo: Hyperkalemic participants were randomized to Placebo for the 9 week double-blind phase.
- HYP Open-Label Dichlorphenamide: Hyperkalemic participants received Dichlorphenamide for the 52 week open-label phase.
- HOP Double-Blind Dichlorphenamide: Hypokalemic participants were randomized to Dichlorphenamide for the 9 week double-blind phase.
- HOP Double-Blind Placebo: Hypokalemic participants were randomized to Placebo for the 9 week double-blind phase.
- HOP Open-Label Dichlorphenamide: Hypokalemic participants received Dichlorphenamide for the 52 week open-label phase.
Arm/Group | HYP Double-Blind Dichlorphenamide | HYP Double-Blind Placebo | HYP Open-Label Dichlorphenamide | HOP Double-Blind Dichlorphenamide | HOP Double-Blind Placebo | HOP Open-Label Dichlorphenamide
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/9 | 0/17 | 0/24 | 1/20 | 3/40
Other Adverse Events (participants affected / at risk) | 9/12 | 3/9 | 12/17 | 20/24 | 11/20 | 32/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HYP Double-Blind Dichlorphenamide (N=12) | HYP Double-Blind Placebo (N=9) | HYP Open-Label Dichlorphenamide (N=17) | HOP Double-Blind Dichlorphenamide (N=24) | HOP Double-Blind Placebo (N=20) | HOP Open-Label Dichlorphenamide (N=40)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Occurred in the pre-treatment screening period.
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HYP Double-Blind Dichlorphenamide (N=12) | HYP Double-Blind Placebo (N=9) | HYP Open-Label Dichlorphenamide (N=17) | HOP Double-Blind Dichlorphenamide (N=24) | HOP Double-Blind Placebo (N=20) | HOP Open-Label Dichlorphenamide (N=40)
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
EYE PAIN (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
PHOTOPSIA (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 1
VISUAL DISTURBANCE (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 2
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
ASTHENIA (General disorders) | 0 | 1 | 1 | 0 | 1 | 1
FATIGUE (General disorders) | 0 | 0 | 1 | 3 | 0 | 4
MALAISE (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
OEDEMA (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
CORNEAL GRAFT REJECTION (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
CYSTITIS ESCHERICHIA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 3
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
TONSILLITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2 | 5
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
ANOREXIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 3
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
COGNITIVE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 5 | 2 | 8
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1
DYSARTHRIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0 | 1 | 4 | 0 | 5
HEADACHE (Nervous system disorders) | 0 | 1 | 1 | 3 | 1 | 3
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 1
LETHARGY (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 2
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 8 | 3 | 9 | 9 | 1 | 12
POLYNEUROPATHY (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 0 | 1 | 2 | 0 | 2
DEPRESSED MOOD (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
NERVOUSNESS (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
NIGHTMARE (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
OILY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 2
FOOT OPERATION (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Sample sizes in the trial were limited by slow recruitment and the trial was concluded before attainment of the target numbers of subjects. Statistical analyses were conducted using smaller group sizes than planned, particularly for HYP subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes